CLINICAL TRIAL: NCT01212172
Title: Side-by-Side Comparison of 810 nm Diode Laser Technology With Low Fluence-High Repetition Rate vs Low Fluence-Vacuum Assist - A Split - Extremity Efficacy , Safety and Tolerability Study
Brief Title: Comparison of Efficacy, Safety and Tolerability of Two Different 810 nm Diode Lasers for Hair Reduction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Christopher Zachary, MBBS, FRCP, University of California, Irvine
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-7704
Record Dates: First submitted 2010-09-22; First posted 2010-09-30 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2015-10

CONDITIONS: Hypertrichosis
Keywords: Hair removal; Laser; Diode laser
MeSH Terms: conditions — Hypertrichosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soprano/SHR (Active Comparator): Alma Soprano/SHR 810 nm Diode Laser
  Interventions: Device: Soprano/SHR
- LightSheer (Active Comparator): LightSheer Duet 810 nm diode laser
  Interventions: Device: LightSheer

INTERVENTIONS:
Device: Soprano/SHR — For the Soprano, the constant motion technique will be used with a fluence ranging between 6 J/cm2 and 10 J/cm2, 10 Hz, 20 ms pulse duration. The constant motion technique involves treating 100 cm2 areas with multiple passes until reaching the cumulative energy dose of 8 kJ. Thus, the hand piece is kept in constant motion to deliver continuous low fluence that will build up energy over time.
  Other Names: Soprano/SHR laser
  Arms: Soprano/SHR
Device: LightSheer — The LightSheer/Duet will be used with conventional single pass (stamping) of the handpiece using settings of single pulse fluence of up to 14 J/cm2 and low vacuum settings.
  Other Names: Duet LightSheer
  Arms: LightSheer

SUMMARY:
The purpose of this research study is to compare two different 810 diode laser systems (Soprano XL (SHR Mode)and Light Sheer Duet) for laser hair removal. The goal is to determine if each laser system is effective at reducing the amount of hair on the lower legs or the axilla (arm pit). Another goal is determine the subject's perspective on the treatment including tolerability and effectiveness.

DETAILED DESCRIPTION:
This side-by-side split body, blinded, randomized single-center study is comparing two different 810 nm diode laser technologies for the purpose of permanent hair reduction to determine the effectiveness and subject's tolerance for hair reduction. Twenty volunteers will be enrolled into this study. Subjects will receive a total of 5 treatments of either axilla or lower legs. 10 patients will have both axilla treated while the other 10 subjects will have the lower legs treated. Placement to the axilla treatment group vs. the lower leg treatment group is random.

Treatment areas will be randomized to receive Soprano SHR treatment or Light Sheer/Duet treatment. One extremity (example: right axilla) will receive Soprano SHR treatment and the contra-lateral extremity (example: left axilla) will receive Duet treatment. The treatments will occur every 6 - 8 weeks and then there will be follow up visits at 1 month, 6 months, and 12 months after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age.
2. Subjects must be in reasonably good health as defined by the Investigator.
3. Subject agrees to avoid tanning during their participation in this trial.
4. Subject has Fitzpatrick skin types I-V and dark brown hair.
5. Subjects must agree to avoid shaving legs less than 72 hours prior to a study visit.
6. Subjects have indicated willingness to participate in the study by signing an informed consent document.

Exclusion Criteria:

1. Subject is pregnant, lactating, or planning to get pregnant within the study period.
2. Subject is unwilling to use birth control during the study period if of child bearing age.
3. Subject has a known history of photosensitivity or use of medication with photosensitizing properties.
4. Subject has skin disease on exam at screening.
5. Subject has history or evidence of any chronic or reoccurring skin disease or disorder(e.g., psoriasis, Netherton syndrome, etc.) affecting the treatment area.
6. Subject has a history of keloid or hypertrophic scar formation.
7. Subject has a tattoo in the treatment area.
8. Subject has been tanning within the past 30 days.
9. Subject has history of confounding cancerous or pre-cancerous skin lesions in the treatment area.
10. Subject has used prohibited therapies (electrolysis, threading, waxing, depilatory), prohibited oral prescription medications (isotretinoin, steroids), or prohibited topical meds (steroids) on the treatment area within 30 days prior to enrollment.
11. Subject is unwilling to discontinue use of above listed prohibitive therapies for the duration of treatment.
12. Subject has a history of laser hair removal in the treatment area.
13. Subject has participated in any clinical trial involving an investigational drug or cosmetic product or procedure within the past 30 days.
14. The investigator feels that for any reason the subject is not eligible to participate in the study.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher B Zachary, MBBS, FRCP, Principal Investigator — University of California, Irvine
Locations (1):
- Department of Dermatology Clinical Research, Irvine, California, United States

REFERENCES:
- See also: UC Irvine Department of Dermatology Clinical Research — http://www.dermatology.uci.edu/clinical_research.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Soprano Duet 810 nm Diode Laser: Soprano Duet 810 nm diode laser
  Soprano/SHR: For the Soprano, the constant motion technique will be used with a fluence ranging between 6 J/cm2 and 10 J/cm2, 10 Hz, 20 ms pulse duration. The constant motion technique involves treating 100 cm2 areas with multiple passes until reaching the cumulative energy dose of 8 kJ. Thus, the hand piece is kept in constant motion to deliver continuous low fluence that will build up energy over time.
- LightSheer Duet 810 nm Diode Laser: Soprano and LightSheer Duet 810 nm diode laser
  LightSheer: The LightSheer/Duet will be used with conventional single pass (stamping) of the handpiece using settings of single pulse fluence of up to 14 J/cm2 and low vacuum settings.
Period: Overall Study
Arm/Group | Soprano Duet 810 nm Diode Laser | LightSheer Duet 810 nm Diode Laser
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Side-by Side Comparsion of Soprano/SHR to Light Sheer: Alma Soprano/SHR 810 nm Diode Laser
  Soprano/SHR: For the Soprano, the constant motion technique will be used with a fluence ranging between 6 J/cm2 and 10 J/cm2, 10 Hz, 20 ms pulse duration. The constant motion technique involves treating 100 cm2 areas with multiple passes until reaching the cumulative energy dose of 8 kJ. Thus, the hand piece is kept in constant motion to deliver continuous low fluence that will build up energy over time.
  LightSheer Duet 810 nm diode laser
  LightSheer: The LightSheer/Duet will be used with conventional single pass (stamping) of the handpiece using settings of single pulse fluence of up to 14 J/cm2 and low vacuum settings.
Arm/Group | Side-by Side Comparsion of Soprano/SHR to Light Sheer
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Hair Growth
Description: % reduction from baseline hair count at time points 1 month, 6 months and 12 months [following last (5th laser) treatment]
Time Frame: 1 month, 6 month, 12 month
Measure: Mean (Standard Deviation); unit: % hair reduction
Arm/Group | Soprano/SHR | LightSheer
Number analyzed (Participants) | 20 | 20
% hair reduction
  1 month | 57.6 (34.03) | 52.1 (32.2)
  6 month | 39.3 (23.3) | 29.9 (21.7)
  12 month | 47.5 (38.41) | 44.7 (43.2)
Statistical Analysis 1: Comparison: Soprano/SHR vs LightSheer; Test type: Superiority or Other; p = 0.2879, t-test, 1 sided; Mean Difference (Final Values) = 7.9, 95% CI 2-sided [-6.7 to 21.1]

2. Secondary Outcome: Pain Rating Scale
Description: Pain during each treatment was measured subjectively by patients on a 0-10 visual analogue scale (0=no pain, 10=unbearable pain).
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: Units on a Scale
Arm/Group | LightSheer | Soprano/SHR
Number analyzed (Participants) | 20 | 20
Units on a Scale | 3.6 [2.8 to 4.5] | 2.7 [1.8 to 3.5]

ADVERSE EVENTS:
Time Frame: At each laser treatment visit and all post-laser treatment follow-up visits (1 month, 6 months, 12 months)
Groups:
- Soprano/SHR 810 nm Diode Laser: Alma Soprano/SHR VS Light Sheer Duet 810 nm Diode Lasers
  Right Axilla or Lower Leg
  Soprano/SHR: For the Soprano, the constant motion technique will be used with a fluence ranging between 6 J/cm2 and 10 J/cm2, 10 Hz, 20 ms pulse duration. The constant motion technique involves treating 100 cm2 areas with multiple passes until reaching the cumulative energy dose of 8 kJ. Thus, the hand piece is kept in constant motion to deliver continuous low fluence that will build up energy over time.
- Light Sheer 810 nm Diode Laser: Light Sheer 810 nm Diode Laser
  Left Axilla or Lower Leg
  LightSheer: The LightSheer/Duet will be used with conventional single pass (stamping) of the handpiece using settings of single pulse fluence of up to 14 J/cm2 and low vacuum settings.
Arm/Group | Soprano/SHR 810 nm Diode Laser | Light Sheer 810 nm Diode Laser
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 6/20 | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soprano/SHR 810 nm Diode Laser (N=20) | Light Sheer 810 nm Diode Laser (N=20)
Burn (General disorders) | 6 (8) | 5 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No